CLINICAL TRIAL: NCT06633640
Title: Evaluation of an Algae-Based Biphasic Bone Graft Material and Collagen Membrane in the Treatment of Periodontal Intrabony Defects: A Randomized Clinical Trial
Brief Title: Evaluation of an Algae-Based Biphasic Bone Graft Material and Collagen Membrane in the Treatment of Periodontal Intrabony Defects
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rahma Omar B. Ahmed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18224
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Intrabony Periodontal Defect; Periodontitis
Keywords: Algae-Based Biphasic Graft substances
MeSH Terms: conditions — Periodontitis | interventions — Algipore

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Conventional flap with algae-based substitute (AlgOss) combined with collagen membrane
  Interventions: Combination Product: Conventional flap with algae-based substitute (AlgOss) combined with collagen membrane.
- Control group (No Intervention): Conventional flap with collagen membrane

INTERVENTIONS:
Combination Product: Conventional flap with algae-based substitute (AlgOss) combined with collagen membrane. — The graft material will be prepared following the manufacturer instruction, transferred into a sterile cup than the mixture is condensed without overfilling in the intrabony defect to the level of the surrounding bony walls. The filled site will be than covered with collagen membrane.
  Arms: Intervention

SUMMARY:
Periodontal diseases are one of the most prevalent chronic diseases involving a spectrum of inflammatory conditions. Intrabony defects, also known "vertical defects," are specific osseous and morphological defects and one of the consequences and end result of periodontitis. Intrabony defects are particularly associated with periodontal progression however certain patient-related factors play important role in its management such as plaque management, smoking, medical history, tooth mobility and endodontic condition.

Periodontal repair is aimed to gain periodontal attachment using various modalities in severely compromised teeth, decrease pocket depth, and stabilize gingival recession. Different types of biomaterial substitutes and bone graft materials are available, but the choice of suitable "golden" type or technique is difficult and dependent on various factors particularly anatomical variations, cost effective, clinical situations, the systemic general condition, operation site, socioeconomic conditions and the surgeon choice.

The current therapeutic options mainly focus on minimize symptoms and prevent disease progression but are not able to fully restore damaged bone and periodontal supporting tissues. Many of these regenerative approaches, (e.g. bone grafts) provided variable and unpredictable clinical outcomes. Therefore, it is imperative to develop alternative regenerative strategies.

There is necessity to introduce novel and alternative materials of natural and synthetic origins for bone grafting use in dental field. This requires well performed clinical trials on humans to understand the effects of such materials (e.g the marine algae-based substitutes and biodegradable (absorbable) materials) either as a single or combined formula.

The aim of the current clinical study is to evaluate the clinical efficacy of an algae-based biphasic bone graft material (AlgOss 20/80) and collagen membrane in the treatment of patient with intrabony periodontal defects.

DETAILED DESCRIPTION:
Study population Recruited patients attending the dental clinic at the faculty of dentistry of the University of Cairo, Egypt will be included following the study eligibility criteria.

Population: Patients with periodontal intrabony defects (Stage III and IV periodontitis).

Intervention: Conventional flap with algae-based substitute (AlgOss) combined with collagen membrane.

Control: Conventional flap with collagen membrane.

Outcomes:

Primary outcome:

- Clinical attachment level (CAL)

Secondary outcomes:

* Bleeding on probing (BOP)
* Plaque index (PI)
* Probing pocket depth (PPD)
* Gingival recession (GR)
* Defect depth and width
* Radiographic depth and width
* Postoperative care and satisfaction assessment

ELIGIBILITY:
Inclusion Criteria:

1. The age is between ≥ 20 to ≤ 65 years old.
2. Presence of intrabony defect
3. Systematically free.
4. The subjects understand the purpose of the study, adhere to the study protocol and given consent to be included in the study.
5. Adequate plaque control and stable periodontal status (full-mouth bleeding score on probing: <25%, and full- mouth plaque score: <25%)

Exclusion Criteria:

1. Smokers
2. Any infection particularly at the intervention site.
3. Teeth mobility more than grade 1.
4. Pregnant or lactating women.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | From date of enrolment until the date of first documented progression i.e.at least12 months after the last enrolment.
  The CAL will be measured from the cementoenamel junction (CEJ) to the base of the sulcus or pocket

SECONDARY OUTCOMES:
Probing pocket depth (PPD) | From date of enrolment until the date of first documented progression i.e.at least12 months after the last enrolment.
  Probing pocket depth (PPD):
  PPD is determined by measuring the distance from the gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.

OTHER OUTCOMES:
Bleeding on probing (BOP) | From date of enrolment until the date of first documented progression i.e.at least12 months after the last enrolment.
  The BOP is the primary parameters to assess gingivitis and recorded using gingival index (GI) score. The GI and gingival bleeding caused by running a Williams periodontal probe inside the pocket on the mesial, distal, buccal, and palatal surfaces of all teeth will be evaluated following. The GI of each individual will be determined by calculating the values determined for each tooth and obtaining the averages.
Plaque index (PI) | From date of enrolment until the date of first documented progression i.e.at least12 months after the last enrolment.
  The PI will be evaluated by probing the mesial, distal, buccal, and palatal surfaces of all teeth using a Williams periodontal probe. The PI of each individual will be determined by summing the values obtained for each tooth and calculating the averages.
Gingival recession (GR) | From date of enrolment until the date of first documented progression i.e.at least12 months after the last enrolment.
  GR is usually recorded as a clinical measure when assessing regenerative outcome as indicators of level of tissue coverage as well as new attachment. It is measured from the CEJ to the most apical extension of the gingival margin using periodontal probe at six sites per tooth.
Depth and width of defect (including Radiographic) | From date of enrolment until the date of first documented progression i.e.at least12 months after the last enrolment.
  Defect depth will be measured as the distance between the alveolar bone crest and the most apical extension of the bone defect. The width of defect will be measured as the horizontal distance between the alveolar bone crest at the intrabony defect in the direction towards the center of the tooth. Radiographic outcomes at base line, 6 ad 12 months will be measured using ImageJ software.
Postoperative care and satisfaction assessment | From date of enrolment until the date of first documented progression i.e.at least12 months after the last enrolment.
  Patients will be followed up for assessment of their satisfaction using a rating scale from 0 (no pain) to 10 (extremely severe pain) .

CONTACTS AND LOCATIONS:
Locations (1):
- Periodontology Clinic, Faculty of Oral and Dental medicine, University of Cairo, Egypt., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paolantonio M. Combined periodontal regenerative technique in human intrabony defects by collagen membranes and anorganic bovine bone. A controlled clinical study. J Periodontol. 2002 Feb;73(2):158-66. doi: 10.1902/jop.2002.73.2.158. PMID 11895280